CLINICAL TRIAL: NCT02871323
Title: A Phase 1, Single Arm, Single Center Pilot Study of Medi4736, an Anti-Pdl1 Therapy, for Patients With Myelofibrosis
Brief Title: Durvalumab in Treating Patients With Primary, Post-Polycythemia Vera, or Post-Essential Thrombocythemia Myelofibrosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decided to withdraw the study after it opened for enrollment but before any patients were enrolled
Sponsor: Northwestern University (Other)
Collaborators: Celgene (Industry); The Leukemia and Lymphoma Society (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16H05; STU00202833 (CTRP (Clinical Trial Reporting Program)); NU 16H05 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-01024 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-08-09; First posted 2016-08-18 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Primary Myelofibrosis
Keywords: Myelofibrosis Transformation in Essential Thrombocythemia
MeSH Terms: conditions — Polycythemia Vera; Primary Myelofibrosis | interventions — durvalumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (durvalumab) (Experimental): Patients receive durvalumab IV over approximately 1 hour on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients with SD, no new inter-current illness, and no unacceptable toxicity, may continue treatment beyond 3 courses.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
The main purpose of this investigational research study is to determine how safe and tolerable the study drug, MEDI4736 (Durvalumab), is in patients with myelofibrosis (MF). The study drug belongs to a group of drugs called immune checkpoint inhibitors, which have shown promise in other forms of cancer, such as melanoma and lung cancer. One of the effects that this drug has is to activate the patient's own natural immune system. The purpose of this study is to examine the safety and tolerability of the study drug, to study how effective it is at treating patients with myelofibrosis, and to explore how certain markers in the patient's blood and/or bone marrow may be affected by the study drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of anti-programmed cell death 1 ligand 1 (PDL1) therapy in patients with myelofibrosis.

SECONDARY OBJECTIVES:

I. Changes in MF symptom burden. II. Changes in spleen size. III. Blood and/or bone marrow samples.

TERTIARY OBJECTIVES:

I. To determine the rate of lymphocyte subset response to anti-PDL1 therapy, as measured by the percent increase in cluster of differentiation (CD)4+CD25+PD-L1+ T-lymphocytes and CD4+CD62L+CD127+ T lymphocytes in post-treatment peripheral blood samples.

II. To characterize changes in the cytokine profile in response to anti-PDL1 therapy.

III. To measure soluble PDL1 by enzyme-linked immunosorbent assay (ELISA) in post-treatment blood and/or bone marrow samples and programmed cell death-1 (PD1)/PDL1 by immunohistochemistry on bone marrow samples and correlate with treatment response.

OUTLINE:

Patients receive durvalumab intravenously (IV) over approximately 1 hour on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease (SD), no new inter-current illness, and no unacceptable toxicity, may continue treatment beyond 3 courses.

Patients will be followed every 3 months for up to two years starting from Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of primary myelofibrosis (PMF), post-polycythemia vera (post-PV) myelofibrosis (MF), or post-essential thrombocythemia (post-ET) MF using World Health Organization Criteria
* Patients must have disease that requires therapy, including intermediate-1, intermediate-2, or high-risk disease according to the International Prognostic Scoring System (IPSS) or Dynamic-IPSS
* Patients must be resistant to, intolerant of, or ineligible for Janus kinase (JAK)2 inhibitor therapy, or have refused such therapy
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined below:
* Absolute neutrophil count >= 1.0 x 10^9/L
* Platelets >= 75 x 10^9/L
* Total bilirubin =< institutional upper limit of normal (ULN) (or =< 3 X ULN if Gilbert's syndrome present or if bilirubin increase related to MF)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase[SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SPGT]) =< 2.5 X institutional ULN
* Creatinine clearance >= 50 mL/min/1.73 m^2 (calculated by estimated glomerular filtration rate [eGFR] from EPIC)
* Female subjects who are pregnant or breast-feeding are not eligible; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; likewise, should a female partner of a male patient become pregnant or suspect she is pregnant while participating in the study, he should inform his treating physician and the female partner should call her physician immediately
* Female of child bearing potential (FOCBP) must have a negative pregnancy test (serum or urine) within 7 days prior to registration on study; NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis, Crohn's disease], diverticulitis with the exception of a prior episode that has resolved or diverticulosis, celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener's syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis, uveitis; etc.) within the past 3 years prior to the start of treatment

  * The following are exceptions to this criterion: subjects with vitiligo or alopecia; subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; or subjects with psoriasis not requiring systemic treatment
* Known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or evidence of active hepatitis B virus (HBV)
* Current or prior use of immunosuppressive medication within 14 days prior to first dose of durvalumab; the following are exceptions to this criterion: intranasal, inhaled, topical or local steroid injections (eg. intra-articular injection); steroids as premedication for hypersensitivity reactions; systemic corticosteroid at physiologic doses not to exceed 10 mg/day of prednisone or equivalent; (NOTE: If systemic corticosteroids are part of the treatment regimen for the indication under study, the systemic corticosteroid is permitted)
* Female subjects who are pregnant, breast-feeding or female patients of reproductive potential who are not employing an effective method of birth control from starting dose of durvalumab (cycle 1 day 1), including dosing interruptions through 90 days after receipt of the last dose of durvalumab are not eligible; female subjects should agree to refrain from egg cell donation while taking durvalumab and for at least 90 days after the last dose of durvalumab
* Male subjects who are not employing an effective method of birth control from starting dose of durvalumab (cycle 1 day 1), including dosing interruptions through 90 days after receipt of the last dose of durvalumab are not eligible; male subjects should agree to refrain from sperm donation while taking durvalumab and for at least 90 days after the last dose of durvalumab; should a female partner of a male patient become pregnant or suspect she is pregnant while participating in the study, he should inform his treating physician and the female partner should call her physician immediately
* History of hypersensitivity to durvalumab or any excipient
* Receipt of live attenuated vaccination within 30 days prior the first dose of durvalumab
* Patients may not be receiving any other investigational agents within 2 weeks prior to registration
* Patients who have had prior exposure to checkpoint blockade therapy, such as anti-PD-1/PD-L1, anti-cytotoxic T-lymphocyte associated protein 4 (CTLA4), anti-CD137, and anti-OX40 antibody therapy, are not eligible
* Patients who have an inter-current illness including, but not limited to any of the following, are not eligible:

  * Severe hypertension that is not controlled on medication (>= 140/90 mmHg for 3 consecutive readings)
  * Ongoing or active infection requiring systemic treatment
  * Congestive heart failure with New York Heart Association (NYHA) classification of 3
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Patients with another malignancy, unless they have been disease free for 3 years prior to registration (with the exception of squamous cell carcinoma or basal cell carcinoma of the skin or cervical intraepithelial neoplasia)
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 2 years
  To determine the safety profile of anti-PDL1 therapy in patients with myelofibrosis, adverse events will be assessed by number, frequency, and severity according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

SECONDARY OUTCOMES:
Changes in MF symptom burden | Baseline up to 2 years
  Changes in MF symptom burden will be assessed using the validated Patient Reported Outcome tool called the Myeloproliferative Neoplasm (MPN)-Symptom Assessment Form (SAF).
Changes in spleen size | Baseline up to 2 years
  Change in spleen size will be assessed by physical examination (palpation) OR ultrasound as part of standard of care.
Response to anti-PDL1 treatment in blood | Up to 2 years
  Response to anti-PDL1 treatment will be defined in accordance with the revised/modified International Working Group (IWG) Response Criteria and will be assessed by blood samples.
Response to anti-PDL1 treatment in bone marrow | Up to 2 years
  Response to anti-PDL1 treatment will be defined in accordance with the revised/modified International Working Group (IWG) Response Criteria and will be assessed by bone marrow samples.

OTHER OUTCOMES:
Rate of lymphocyte subset response to anti-PDL1 therapy | Up to 84 days
  Determine the rate of lymphocyte subset response to anti-PDL1 therapy as measured by the percent increase in lymphocytes in post-treatment peripheral blood samples.
Change in the cytokine profile in response to anti-PDL1 therapy | Up to 84 days
  Blood samples will be used to assess any change in the cytokine profile in response to anti-PDL1 therapy.
Change in protein expression in response to anti-PDL1 therapy | Up to 84 days
  To measure soluble PDL1 by ELISA in post-treatment blood and/or bone marrow samples along with PD1/PDL1 by immunohistochemistry on bone marrow samples and correlate both with treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Brady Stein, MD, MHS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States